CLINICAL TRIAL: NCT06753045
Title: Health Electronic Assessment of Risks and Trends Using Biometric Equipment and Technology: HEARTBEAT
Brief Title: Health Electronic Assessment of Risks and Trends Using Biometric Equipment and Technology
Acronym: HEARTBEAT
Status: Recruiting | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-652
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Heart Diseases
Keywords: Heart failure; Coronary artery disease; Stroke/TIA; Diabetes mellitus; Chronic kidney disease; Cardiac arrhythmias; Smart watch; Atrial fibrillation; A-fib; Artificial intelligence; Machine learning
MeSH Terms: conditions — Heart Diseases; Heart Failure; Coronary Artery Disease; Diabetes Mellitus; Renal Insufficiency, Chronic; Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort arm: Patients with at least one cardiovascular disease, 9500 subjects.
  Interventions: Other: Smartwatch
- Healthy arm: Patients visiting a primary care provider for any reason without any cardiovascular diseases, 500 subjects.
  Interventions: Other: Smartwatch

INTERVENTIONS:
Other: Smartwatch — Sensors on the smartwatch will measure vitals such as heart rate, blood pressure, oxygen saturation, body composition, and electrocardio gram (ECG)

SUMMARY:
This is a phase 0, non-interventional, longitudinal, electronic data capture (EDC) study to facilitate the HEARTBEAT Study project has set out to explore the potential use of smartwatches in collecting and analyzing biometric data to improve the detection, identification, and understanding of cardiovascular diseases and related conditions by SAMSUNG and Tulane. The study will include up to ten thousand adult subjects tasked with wearing a smartwatch to collect digital biomarker data over a 1 year period. Concurrent to smartwatch data collection, subjects will be instructed to complete questionnaires via the Huma Decentralized Clinical Trials (HUMADCT) platform. There are no investigational drugs or interventions administered as part of this study.

DETAILED DESCRIPTION:
The central hypothesis in the HEARTBEAT project posits that cardiovascular events are preceded by abnormalities in biometric signals obtained from a smartwatch. These abnormalities may include, but are not limited to, patterns of heart rate, heart rate variability, oxygen saturation, as well as raw PPG signals. By leveraging advanced analytics and machine learning algorithms on smartwatch-derived biometric data, the investigators plan to identify patterns and markers that signal an increased cardiovascular disease risk.

The study will use an end-to-end decentralized approach for data collection. Huma and Alcedis, the electronic data capture (EDC) agencies, will act as the data storage facilitator for 10,000 eligible subjects. The Principal Investigators (PIs) and trained site staff members will assess healthy subjects based on their clinical opinion. If the subjects meet the eligibility criteria and are interested in participating, they will be consented by Tulane.

During the study enrollment phase, a smartwatch will be provided to the subjects, who will then be trained on the study procedures, the web-based questionnaire, and the use of the wearable device. The subjects will be asked to wear the device for one year, after which they will return it to Tulane.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one cardiovascular disease (heart failure, cardiac arrhythmias, chronic kidney disease, coronary artery disease, history of stroke/Transient Ischemic Attack (TIA), or diabetes mellitus).
* Patients visiting a primary care provider for any reason without any of the previously mentioned cardiovascular diseases. (Healthy cohort, limited up to 500 patients throughout the study).

Exclusion Criteria:

* Participants who cannot read, speak, and/or understand English.
* Participants with cognitive impairments who are unable to give informed consent or sign their HIPAA form.
* Participants with cognitive impairments affecting their ability to be compliant with wearing and maintaining wearable devices.
* Participants who are pregnant.
* Participants with tattoos, scars, or skin adhesions that would not allow for Photoplethysmography (PPG) recordings to be collected from a wrist-worn device.
* Participants with neurological disorders that may interfere with device signal quality (e.g., hand tremors).
* Participants with a pacemaker.
* Participants with allergies to watch and/or wristband materials.
* Participants with known plans to permanently leave the state of Louisiana within the observational period.
* Participants who have no known medical history with any of the enrolling institutions.
* Patients without a compatible smartphone (iOS 13 & Android 11 at minimum).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 10,000 patients older than 18 years who will either be healthy or with a pre-existing heart condition.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of cardiovascular events indicative of progression of pre-existing cardiovascular conditions | 1 Year
  These endpoints will be collected from the electronic health records using the International Classification of Diseases Tenth Edition (ICD-10) codes, prompted by a patient survey conducted via the use of a smart phone app. The investigators will use the the patient's survey answers as a prompt to check the EMR. If in the survey a patient mentions they had a cardiovascular incidence, then the EMR data will be checked to see the reports from the ER visit to confirm the incidence. The number that will be reported is the total number of cardiovascular incidences in each patient over the period of 1 year.
The incidence of new cardiovascular diseases events | 1 Year
  These endpoints will be collected from the electronic health records using the International Classification of Diseases Tenth Edition (ICD-10) codes, prompted by a patient survey conducted via the use of a smart phone app. The investigators will use the the patient's survey answers as a prompt to check the EMR. If in the survey a patient mentions they had a cardiovascular incidence, then the EMR data will be checked to see the reports from the ER visit to confirm the incidence and check to confirm if the patient developed a new cardiovascular disease. The number that will be reported is the total number of cardiovascular incidences in each patient over the period of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane University
Locations (3):
- United States (3):
  - East Jefferson General Hospital, New Orleans, Louisiana
  - Tulane University Medical Group Clinics, New Orleans, Louisiana
  - University Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No